CLINICAL TRIAL: NCT01333280
Title: Efficacy of Dual Focus Mutual Aid for Persons With Co-occurring Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Michigan University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephen Magura, Director, Evaluation Center, Western Michigan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUALFOCUSAID; 1R01DA023119-01A1 (NIH)
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Substance Abuse; Mental Disorders
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders | interventions — Salvage Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double Trouble (DTR) group (Experimental): Double Trouble in Recovery groups
  Interventions: Behavioral: Double Trouble in Recovery
- Treatment as usual (Active Comparator): Treatment as usual while on a waiting list for DTR groups
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Double Trouble in Recovery — DTR is a 12 Step-based fellowship for individuals with co-occurring problems of substance abuse and mental illness
  Other Names: 12 Step groups
  Arms: Double Trouble (DTR) group
Behavioral: Treatment as usual — Receive usual treatment at the programs
  Arms: Treatment as usual

SUMMARY:
The purpose of the study is to determine whether adding "dual focus" mutual aid groups to formal treatment for people dually diagnosed with substance abuse and mental illness is effective in improving treatment outcomes.

NO VOLUNTEERS ARE ACCEPTED. ENROLLMENT IS LIMITED TO CLIENTS OF THE PARTICIPATING TREATMENT PROGRAMS.

DETAILED DESCRIPTION:
This study builds on two previous studies by the principal investigator, which found that participation in an established and growing "dual-focus" mutual aid model (Double Trouble in Recovery; DTR) by persons with co-occurring substance use and psychiatric disorders was associated with drug/alcohol abstinence and improved psychiatric outcomes. However, these findings are limited as they are based on studies using an observational design with existing DTR groups and a pre-post design with a historical control. This new application seeks to confirm and significantly extend this research by conducting a randomized clinical trial (RCT) of DTR at multiple treatment sites.

The specific study aims are:

1. To conduct a multi-site RCT to determine the efficacy of "dual focus" 12-step mutual aid groups for persons with co-occurring substance use and mental disorders. Substance-using patients who are admitted to psychiatric outpatient clinics will be randomly assigned within each clinic to (i) DTR group participation plus standard treatment, or (ii) standard treatment as usual (wait list for DTR). The primary outcome is drug/alcohol use. The secondary outcomes are psychiatric medication adherence; quality of life; treatment retention; and traditional 12 step group participation. Major assessments will occur at baseline and 6 months later.
2. To determine the therapeutic mechanisms mediating between DTR participation and behavioral outcomes. Hypothesized mediating variables will include both "common process" factors across treatments, e.g., coping, self-efficacy and social support; and factors relatively unique to mutual aid, e.g., mutual aid group processes, 12-step attitudes and spirituality.
3. To determine the personal, social/environmental and treatment-related variables which predict DTR affiliation.
4. To describe the development of DTR groups and the conditions needed to sustain them.

Federal substance abuse and mental health policy encourages the use of evidence-based interventions, yet rigorous evaluation data are scant for mutual aid groups. In particular, this research will lead to recommendations for improving the integration of formal treatment with mutual aid for persons with co-occurring disorders. Moreover, by conducting the proposed RCT, the study will substantially raise the standard by which mutual aid is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* admission to one of the participating treatment programs
* substance abuse/dependence
* 18-65 years of age

NO VOLUNTEERS ARE ACCEPTED. ENROLLMENT IS LIMITED TO CLIENTS OF THE THE PARTICIPATING TREATMENT PROGRAMS.

Exclusion Criteria:

* Inability to conduct an interview in English or participate in English- language DTR groups
* Appears intoxicated on drugs or alcohol
* Carries a diagnosis of mental retardation
* Deemed actively psychotic by the clinic's intake coordinator
* Appears unable to understand and give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2008-07; Primary Completion 2012-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Substance abuse | Study intake and six month follow-up
  Self-reported substance use and saliva toxicology for drugs

SECONDARY OUTCOMES:
psychiatric medication adherence | six month follow-up
  Self-reported adherence to prescribed medications
Traditional 12-step meeting participation | six month follow-up
Treatment retention | six month follow-up
Quality of life | six month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Magura, Ph.D., Principal Investigator — Western Michigan University
Locations (4):
- United States (4):
  - Proaction Health Alliance, Grand Rapids, Michigan
  - Coney Island Hospital, Brooklyn, New York
  - BRC, New York, New York
  - South Beach Psychiatric Center, New York, New York

REFERENCES:
- [Result] Rosenblum A, Matusow H, Fong C, Vogel H, Uttaro T, Moore TL, Magura S. Efficacy of dual focus mutual aid for persons with mental illness and substance misuse. Drug Alcohol Depend. 2014 Feb 1;135:78-87. doi: 10.1016/j.drugalcdep.2013.11.012. Epub 2013 Nov 18. PMID 24342419
- [Result] Matusow H, Guarino H, Rosenblum A, Vogel H, Uttaro T, Khabir S, Rini M, Moore T, Magura S. Consumers' Experiences in Dual Focus Mutual Aid for Co-occurring Substance Use and Mental Health Disorders. Subst Abuse. 2013;7:39-47. doi: 10.4137/SART.S11006. Epub 2013 Mar 6. PMID 23515888
- [Result] Magura S, Mateu PF, Rosenblum A, Matusow H, Fong C. Risk factors for medication non-adherence among psychiatric patients with substance misuse histories. Ment Health Subst Use. 2014 Nov;7(4):381-390. doi: 10.1080/17523281.2013.839574. PMID 25309623
- [Result] Matusow H, Rosenblum A, Fong C, Laudet A, Uttaro T, Magura S. Factors associated with mental health clinicians' referrals to 12-Step groups. J Addict Dis. 2012;31(3):303-12. doi: 10.1080/10550887.2012.694605. PMID 22873191